CLINICAL TRIAL: NCT05781815
Title: Treatment Of Unstable Trochanteric Fracture: A Comparative Study Between DHS And DHS With Trochanteric Stabilization Plate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abdelaleem, resident doctor at orthopaedic department, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-23-02-02
Record Dates: First submitted 2023-03-12; First posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Trochanteric Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DHS (Active Comparator): patients with trochanteric fracture treated with DHS
  Interventions: Procedure: dynamic hip screw
- DHS with Trochanteric stabilizing plate (Active Comparator): patients with trochanteric fracture treated with DHS with trochanteric stabilizing plate
  Interventions: Procedure: dynamic hip screw

INTERVENTIONS:
Procedure: dynamic hip screw — using dynamic hip screw in treatment of trochanteric fracture and dynamic hip screw with trochanteric stabilizing plate

SUMMARY:
compare the results in treatment of unstable trochanteric fracture by using DHS and DHS with Trochanteric Stabilizing plate as regard shaft medialization.neck shaft angle measurment and shaft migration

ELIGIBILITY:
Inclusion Criteria:

* pateints with comminution of medial femoral cortex and loss of continuity of lesser trochanter

Exclusion Criteria:

* stable trochanteric fracture subtrochanteric extension reverse oblique trochanteric fracture

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02-10 (Actual); Primary Completion 2023-08-08 (Estimated); Study Completion 2023-08-08 (Estimated)

PRIMARY OUTCOMES:
neck shaft angle measurment .Harris hip score | 6 months
  measurment of neck shaft angle between two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Babhulkar S. Unstable trochanteric fractures: Issues and avoiding pitfalls. Injury. 2017 Apr;48(4):803-818. doi: 10.1016/j.injury.2017.02.022. Epub 2017 Feb 27. PMID 28284469
- [Background] Ahrengart L, Tornkvist H, Fornander P, Thorngren KG, Pasanen L, Wahlstrom P, Honkonen S, Lindgren U. A randomized study of the compression hip screw and Gamma nail in 426 fractures. Clin Orthop Relat Res. 2002 Aug;(401):209-22. doi: 10.1097/00003086-200208000-00024. PMID 12151898
- [Background] SCHUMPELICK W, JANTZEN PM. A new principle in the operative treatment of trochanteric fractures of the femur. J Bone Joint Surg Am. 1955 Jul;37-A(4):693-8. No abstract available. PMID 13242603
- [Background] Harris WH. Traumatic arthritis of the hip after dislocation and acetabular fractures: treatment by mold arthroplasty. An end-result study using a new method of result evaluation. J Bone Joint Surg Am. 1969 Jun;51(4):737-55. No abstract available. PMID 5783851